CLINICAL TRIAL: NCT07087860
Title: MC220503 Randomized Phase II Rescuing Cancer Immunotherapy With Plasma Exchange in Bladder Cancer 1 (ReCIPE-B1)
Brief Title: Therapeutic Plasma Exchange With Enfortumab Vedotin and Pembrolizumab for Treatment of Bladder Cancers
Acronym: RECIPE-B1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC220503; NCI-2025-04887 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-006413 (Other: Mayo Clinic Institutional Review Board); MC220503 (Other: Mayo Clinic)
Record Dates: First submitted 2025-07-16; First posted 2025-07-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis and Ureter Urothelial Carcinoma; Refractory Bladder Urothelial Carcinoma; Refractory Renal Pelvis and Ureter Urothelial Carcinoma; Stage IV Bladder Cancer AJCC v7; Stage IV Renal Pelvis and Ureter Cancer AJCC v7
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Central Venous Catheters; enfortumab vedotin; Magnetic Resonance Spectroscopy; pembrolizumab; Plasmapheresis; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (TPE, EV, pembrolizumab) (Experimental): Patients undergo TPE via venous access or central line on days 1-3 of cycles 1-3 and receive enfortumab vedotin IV over 30 minutes on days 3 and 10 of cycles 1-3 and on days 1 and 8 of cycle 4 and beyond and pembrolizumab IV over 30 minutes on day 3 of cycles 1-3 and day 1 of cycles 4 and beyond. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI and collection of blood and urine samples throughout the study. Patients may undergo central line placement prior to TPE.
  Interventions: Procedure: Biospecimen Collection; Procedure: Central Venous Cannula Insertion; Procedure: Computed Tomography; Drug: Enfortumab Vedotin; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Plasmapheresis; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Group B (standard of care) (Active Comparator): Patients receive physician's choice of standard of care next-line therapy. Patients also undergo CT, PET/CT, or MRI and collection of blood and urine samples throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Cohort C (TPE, ADC) (Experimental): Patients undergo TPE via venous access or central line on days 1-3 of cycles 1-3 only and receive physician's choice of standard of care ADC IV on day 3 of cycles 1-3 and on day 1 of cycles 4 and beyond. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI and collection of blood and urine samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Central Venous Cannula Insertion; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Plasmapheresis; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Biological: Antibody-Drug Conjugate Therapy

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group B (standard of care)
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Central Venous Cannula Insertion — Undergo central line placement
  Other Names: Central venous catheter; Central Venous Catheter Placement
  Arms: Cohort C (TPE, ADC); Group A (TPE, EV, pembrolizumab)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
  Arms: Cohort C (TPE, ADC); Group A (TPE, EV, pembrolizumab)
Drug: Enfortumab Vedotin — Given IV
  Other Names: AGS 22ME; AGS-22M6E; Anti-Nectin 4 ADC ASG-22CE; Anti-nectin-4 Monoclonal Antibody-Drug Conjugate AGS-22M6E; ASG 22CE; ASG-22CE; ASG22CE; Enfortumab Vedotin-ejfv; Padcev
  Arms: Group A (TPE, EV, pembrolizumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Group A (TPE, EV, pembrolizumab)
Procedure: Plasmapheresis — Undergo TPE
  Other Names: Plasma Exchange; Therapeutic Plasma Exchange; Therapeutic Plasmapheresis
  Arms: Cohort C (TPE, ADC); Group A (TPE, EV, pembrolizumab)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Biological: Antibody-Drug Conjugate Therapy — Given IV
  Arms: Cohort C (TPE, ADC)

SUMMARY:
This phase II trial compares therapeutic plasma exchange followed by enfortumab vedotin and pembrolizumab to standard of care next-line therapy for the treatment of patients with bladder or upper urinary tract cancers that have spread from where they first started (primary site) to other places in the body (metastatic) and that have not responded to previous treatment (refractory). TPE is a process that slowly removes a patient's blood through an intravenous or central line. The blood is sent through a machine that separates the plasma (the liquid part of blood) from other blood components (red cells, white cells, platelets). The plasma is then removed. The remaining blood components are combined with replacement fluid and returned to the patient's bloodstream through the intravenous or central line. Enfortumab vedotin is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of cancer cells. Enfortumab attaches to a protein called nectin-4 on cancer cells in a targeted way and delivers vedotin to kill them. It is a type of antibody-drug conjugate. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Treatment with enfortumab vedotin and pembrolizumab is already approved by the Food and Drug Administration for the treatment of bladder cancer, but TPE is not. Combining TPE with enfortumab vedotin and pembrolizumab may work better than standard of care options for treating metastatic and refractory bladder and urinary tract cancers. This study also evaluates the effect of TPE with standard of care antibody drug conjugates (ADCs) in treating patients with refractory metastatic bladder cancer. ADC therapy is treatment with a monoclonal antibody linked to a chemotherapy drug. It is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of tumor cells, and delivers chemotherapy to kill them. Giving TPE with standard of care ADC therapy may be effective in treating patients with refractory metastatic bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the response rate (overall response rate [ORR]) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 among patients with metastatic bladder cancer (mBCa) who receive therapeutic plasma exchange (TPE) and antibody drug conjugate/immune checkpoint inhibition (ADC/ICI) re-challenge (group A) versus next-line standard of care therapy (group B) after progression on enfortumab vedotin combined with pembrolizumab (EV/pembro). (ReCIPE-B1 [Groups A and B]) II. To evaluate the response rate (ORR) by RECIST version 1.1 among patients with metastatic bladder cancer (mBCa) who receive therapeutic plasma exchange (TPE) and antibody drug conjugate (ADC) re-challenge (Cohort C) versus historical controls after progression on ADC. (CAKE ReCIPE [Cohort C])

SECONDARY OBJECTIVES:

I. To evaluate and compare the overall survival (OS) of patients receiving TPE and ADC/ICI re-challenge versus next-line standard of care. (ReCIPE-B1 [Groups A and B]) II. To evaluate and compare the duration of response (DOR) by RECIST 1.1 between the arms. (ReCIPE-B1 [Groups A and B]) III. To evaluate and compare progression-free survival (PFS) by RECIST 1.1 between the arms. (ReCIPE-B1 [Groups A and B]) IV. To evaluate safety as assessed per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in both treatment arms. (ReCIPE-B1 [Groups A and B]) V. To evaluate patients' quality of life (QoL) among both treatment arms as assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy Induced Peripheral Neuropathy 20 (EORTC QLQ-CIPN20) at baseline and every 12 weeks. (ReCIPE-B1 [Groups A and B]) VI. To evaluate the overall survival (OS) of patients receiving TPE and ADC re- challenge. (CAKE ReCIPE [Cohort C]) VII. To evaluate the duration of response (DOR) by RECIST 1.1. (CAKE ReCIPE [Cohort C]) VIII. To evaluate progression-free survival (PFS) by RECIST 1.1. (CAKE ReCIPE [Cohort C]) IX. To evaluate safety as assessed per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. (CAKE ReCIPE [Cohort C]) X. To evaluate patients' quality of life (QoL) as assessed by EORTC QLQ-CIPN20 at baseline and every 12 weeks. (CAKE ReCIPE [Cohort C])

CORRELATIVE OBJECTIVE:

I. To use circulating exosomes, circulating tumor deoxyribonucleic acid (DNA), and urine tumor DNA for identifying predictive biomarkers of response, progression, or relapse.

OUTLINE: Patients are randomized to 1 of 2 groups. Patients are assigned to Cohort C.

GROUP A: Patients undergo TPE via venous access or central line on days 1-3 of cycles 1-3 and receive enfortumab vedotin intravenously (IV) over 30 minutes on days 3 and 10 of cycles 1-3 and on days 1 and 8 of cycle 4 and beyond and pembrolizumab IV over 30 minutes on day 3 of cycles 1-3 and day 1 of cycles 4 and beyond. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) and collection of blood and urine samples throughout the study. Patients may undergo central line placement prior to TPE.

GROUP B: Patients receive physician's choice of standard of care next-line therapy. Patients also undergo CT, PET/CT, or MRI and collection of blood and urine samples throughout the study.

COHORT C: Patients undergo TPE via venous access or central line on days 1-3 of cycles 1-3 only and receive physician's choice of standard of care ADC IV on day 3 of cycles 1-3 and on day 1 of cycles 4 and beyond. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI and collection of blood and urine samples throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* GROPUS A and B (reCIPE-B1): Histologically proven urothelial carcinoma [American Joint Committee on Cancer (AJCC) 2017] of the bladder (BCa) or upper urothelial tract (UTUC), that has progressed despite enfortumab vedotin and pembrolizumab treatment

  * NOTE: Primary or secondary progression are allowed, therapies are not required to be concurrent or immediately antecedent to enrollment)
* COHORT C (CAKE ReCIPE): Histologically proven urothelial carcinoma (AJCC 2017) of the bladder (BCa) or upper urothelial tract (UTUC), that has progressed despite ADC AND is otherwise not a candidate for Groups A and B

  * NOTE: Patients in Groups A and B who have progressed on that treatment are candidates for this cohort. Such patients must be re-consented and re- enrolled
* Measurable disease per RECIST version (v)1.1
* Eastern Cooperative Oncology Group (ECOG) performance status grade 0, 1, or 2
* Hemoglobin > 7.0 g/dL (obtained ≤ 30 days prior to registration)
* Platelet count ≥ 75,000/mm^3 (obtained ≤ 30 days prior to registration)
* Alanine aminotransferase (ALT) OR aspartate transaminase (AST) ≤ 3.5 x upper limit of normal (ULN) OR total bilirubin ≤ 3 x ULN OR direct bilirubin ≤ 3 x ULN (obtained ≤ 30 days prior to registration)
* Estimated glomerular filtration rate (GFR) ≥ 15 ml/min (obtained ≤ 30 days prior to registration)
* Negative pregnancy test ≤ 8 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to undergo treatment as assigned (group A: TPE + EV/pembro; OR group B: next line standard of care; OR Cohort C TPE + ADC)
* Willingness to provide mandatory blood and fluid specimens for correlative research
* Willingness to provide tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Any of the following histologic variants/divergent differentiation: Any amount of neuroendocrine, micropapillary, or signet ring cell features
* Active malignancies (i.e., progressing or requiring treatment change ≤ 24 months before registration) other than the disease being treated under study

  * EXCEPTIONS:

    * Skin cancer (melanoma or non-melanoma) that is considered completely cured
    * Non-invasive cervical cancer that is considered completely cured
    * Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ considered to have a very low risk of recurrence
    * Localized prostate cancer (T1c/T2N0M0):

      * Gleason score 6, treated by either surgery or ablation ≤ 24 months prior to registration or untreated and under active surveillance
      * Gleason score 3+4 that has been treated (may include surgery or ablation) ≤ 24 months prior to registration and considered to have a very low risk of recurrence (i.e., cT1c or pT2 on prostatectomy specimen)
* History of uncontrolled cardiovascular disease including any of the following ≤ 6 months prior to registration:

  * Significant cardiovascular disease [New York Heart Association (NYHA) class ≥ III], symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction, ventricular fibrillation, Torsades de Pointes, cerebrovascular accident, or transient ischemic attack
  * Psychiatric illness/social situations (e.g., substance abuse) that would limit compliance with study requirements
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participants (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-08-07 (Estimated); Study Completion 2028-08-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (Groups A and B) | Up to 6 months
  ORR is defined as proportion of evaluable patients with complete response (CR) or partial response (PR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
ORR (Cohort C) | Up to 6 months
  ORR is defined as proportion of evaluable patients with complete response (CR) or partial response (PR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) (Groups A and B) | Up to 5 years
  Duration of response is defined as the time from date of objective response (CR or PR) to date of progression per RECIST 1.1 or death due to all causes, whichever occurs first.
DOR (Cohort C) | Up to 5 years
  Duration of response is defined as the time from date of objective response (CR or PR) to date of progression per RECIST 1.1 or death due to all causes, whichever occurs first.
Overall survival (OS) (Groups A and B) | Up to 5 years
  OS is defined as the time from the date of randomization to the date of death due to all causes.
OS (Cohort C) | Up to 5 years
  OS is defined as the time from the date of randomization to the date of death due to all causes.
Progression-free survival (PFS) (Groups A and B) | Up to 5 years
  PFS is defined as the time from the date of study randomization (assignment to study arm) to the date of death due to all causes or disease progression per RECIST 1.1.
PFS (Cohort C) | Up to 5 years
  PFS is defined as the time from the date of study randomization (assignment to study arm) to the date of death due to all causes or disease progression per RECIST 1.1.
Incidence of adverse events (AEs) (Groups A and B) | Up to 5 years
  AEs will be assessed per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of AEs (Cohort C) | Up to 5 years
  AEs will be assessed per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life - EORTC QLQ-CIPN20 (Groups A and B) | Baseline; every 12 weeks (every 4 cycles) until treatment completion, up to 5 years
  Quality of life will be measured by change in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Chemotherapy Induced Peripheral Neuropathy 20 (QLQ-CIPN20) scores, a 20-item questionnaire used to assess the severity of neuropathy symptoms experienced by cancer patients during the past week. Questions are answered on a scale of 1-4 where 1=not at all, 2= a little, 3=quite a bit, and 4=very much. Higher scores indicate greater severity of symptoms.
Quality of life - EORTC QLQ-CIPN20 (Cohort C) | Baseline; every 12 weeks (every 4 cycles) until treatment completion, up to 5 years
  Quality of life will be measured by change in EORTC QLQ-CIPN20 scores, a 20-item questionnaire used to assess the severity of neuropathy symptoms experienced by cancer patients during the past week. Questions are answered on a scale of 1-4 where 1=not at all, 2= a little, 3=quite a bit, and 4=very much. Higher scores indicate greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J. Orme, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials